CLINICAL TRIAL: NCT04031014
Title: High Intensity Focused Electromagnetic Field Device for Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Urogynecology Associates (Other)
Responsible Party: Principal Investigator, William D. Winkelman, Division Director, Boston Urogynecology Associates
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 021-2019
Record Dates: First submitted 2019-07-19; First posted 2019-07-24 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Stress Urinary Incontinence; Urge Incontinence; Urge and Stress; Overactive Bladder
Keywords: Stress urinary incontinence, urge urinary incontinence, overactive bladder
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence, Urge; Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: Active and sham arms 1:1 run in parallel
Who Masked: Participant, Care Provider, Investigator
Masking Description: Two blinded protocols are available on the device, neither investigators, participants or care providers will know the active treatment arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active treatment (Experimental): Treatment with the active treatment protocol of the BTL EMSELLA device twice per week for six treatments total
  Interventions: Device: BTL EMSELLA Active treatment
- Sham treatment (Sham Comparator): Treatment with the sham protocol of the BTL EMSELLA device twice per week for six treatments total
  Interventions: Device: BTL EMSELLA Sham Treatment

INTERVENTIONS:
Device: BTL EMSELLA Active treatment — BTL EMSELLA delivers high intensity focused electromagnetic technology to induce pelvic floor muscle contractions up to maximum intensity of 100% for active treatment
  Arms: Active treatment
Device: BTL EMSELLA Sham Treatment — BTL EMSELLA delivers high intensity focused electromagnetic technology to induce pelvic floor muscle contractions up to maximum intensity of 5% for sham treatment
  Arms: Sham treatment

SUMMARY:
High intensity focused electromagnetic (HIFEM) technology induces deep pelvic floor muscle contractions designed to deliver the equivalent of 11,200 Kegel exercise over 28 minutes, with the intention of increasing neuromuscular tone of the pelvic floor. This study will have looking at treatment of the two of the most common pelvic floor disorders: stress or stress predominant urinary incontinence and urge or urge predominant urinary incontinence.

DETAILED DESCRIPTION:
Pelvic floor dysfunction is common and can include symptoms of urinary incontinence, fecal incontinence and prolapse. Studies suggest that pelvic floor dysfunction may affect up to 25% of women in the United States including 17.1% of women with moderate to severe urinary. While most causes of stress/stress predominant urinary incontinence and urge/urge predominant urinary incontinence are due to of poor pelvic floor musculature and abnormal neuromuscular control, the cause of these abnormalities is not known. Traumatic injuries to the pelvic area, such as in an accident, and complications from vaginal childbirth can contribute to this condition. Some cases are due to a learned behavior (repeated actions of straining).

For most pelvic floor disorders, first line therapy involves behavioral modifications and pelvic floor physical therapy. Physical therapy has proven benefits for treatment of pelvic floor disorders and may improve symptoms in up to 70% of patients with any urinary incontinence (either OAB or SUI), and 60-70% patients with FI. Unfortunately, not all patients are able or willing to undergo treatment with pelvic floor physical therapy. During therapy, patients are undressed, and the therapist works internally palpating the muscles in the vagina and rectum to facilitate rehabilitation. Treatment with the BTL EMSELLA allows for similar rehabilitation of the pelvic floor while patients remain comfortably clothed.

The use of magnetic stimulation to treat pelvic floor disorders has been studied previously. In one prospective cohort study of 91 women, treatment with weekly sessions of perineal magnetic stimulation was associated with improved quality of life and decreased urinary leakage episodes. Magnetic stimulation has also been shown to improve urodynamic parameters, both increasing the maximum urethral pressure for patients with stress incontinence, and increase bladder capacity for those with urgency incontinence. The BTL EMSELLA is a device cleared by the Food and Drug Administration (FDA) for entirely non-invasive electromagnetic stimulation of pelvic floor musculature for the purpose of rehabilitation of weak pelvic muscles and restoration of neuromuscular control for the treatment of male and female urinary incontinence. High intensity focused electromagnetic (HIFEM) technology induces deep pelvic floor muscle contractions designed to deliver the equivalent of 11,200 Kegel exercise over 28 minutes, with the intention of increasing neuromuscular tone of the pelvic floor. This study will look at treatment of the two of the most common pelvic floor disorders: stress or stress predominant urinary incontinence and urge or urge predominant urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

1. Subject provides written informed consent and HIPAA authorization before any study procedures are conducted
2. Age greater than 18
3. Subject has a body mass index (BMI) < 37 kg/m2
4. Subject has stress urinary incontinence, urge incontinence, or mixed urinary incontinence as determined by the QUID;
5. Subject is willing to continue level of core exercise currently being performed or not performed during the study (e.g. gym, Pilates, yoga);
6. Subject is willing to maintain her current prescription and over the counter medications throughout the study without changing them;
7. Subject agrees to comply with the study procedures and visits.

Exclusion Criteria:

1. Subject has used the BTL EMSELLA device previously;
2. Subject has any significant pelvic organ prolapse; stage III or greater
3. Subject is unwilling to maintain current level of exercise throughout the study;
4. Subject planning to have surgery during the study;
5. Subject has untreated malignancy;
6. Subject is pregnant, planning to get pregnant or within 3 months postpartum;
7. Subject has a pacemaker;
8. Subject has and implant or IUD containing metal;
9. Subject has piercing between the waist and knees and is not willing to remove it before each treatment;
10. Subject is using a pessary or other anti-incontinence device
11. Subject has implanted defibrillator, implanted neurostimulator
12. Subject has metal implants
13. Subject has a drug pump

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Patient global impression of improvement (PGI-I) | Baseline, 2 weeks after treatment, 3 months after treatment
  The PGI comprises two companion one-item measures evaluating the following: (a) severity of psychopathology from 1 to 7 and (b) change from the initiation of treatment on a similar seven-point scale. The Patient Global Impression of Improvement (PGI-I) has been validated for use in female patients with urinary incontinence and prolapse. Using this measure we hope to assess for overall improvement in symptoms after treatment. Change from baseline will range from -6 to +6 with higher scores representing better outcomes.

SECONDARY OUTCOMES:
24 hour voiding diary | Baseline, 2 weeks after treatment, 3 months after treatment
  A three-day voiding diary is a validated measure based on the International Consultation on Incontinence Questionnaires and involves measurement of fluid intake, leakage episodes and pad useage. There is high correlation between a 24 hour voiding diary and a 3 day voiding diary with higher rates of compliance. Participants will therefore complete a 24 hour voiding diary prior to enrollment, at the conclusion of treatment and again at a 3 month follow up visit. In addition, patients will answer questions on the frequency of pad use. Using the voiding diary we will look specifically at leakage episodes, urgency episodes.
FSFI | Baseline, 2 weeks after treatment, 3 months after treatment
  The FSFI was developed to measure female sexual function. The FSFI is a 19-item patient-reported outcome measure (PROM), consisting of 6 separate domains of female sexual function, namely desire (items 1-2), arousal (3-6), lubrication (7-10), orgasm (11-13), satisfaction (14-16), and pain (17-19). We will assess for change in total score of the FSFI from pre-treatment to follow up visits. Scores range from 2 to 36 with higher results representing better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Urogynecology Associates, Cambridge, Massachusetts, United States